CLINICAL TRIAL: NCT01493050
Title: Multi-Center Study of the Effect of Sevelamer Carbonate (Renvela®) on Metabolic/Inflammatory/ROS in Diabetics With Nephropathy
Brief Title: The Effects of Sevelamer Carbonate on Diabetic Nephropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gary Striker (Other)
Responsible Party: Sponsor-Investigator, Gary Striker, Principal Investigator, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 11-0973
Record Dates: First submitted 2011-12-13; First posted 2011-12-15 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Diabetic Nephropathy
Keywords: Diabetic Nephropathy; Sevelamer Carbonate
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Sevelamer; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sevelamer Carbonate (Experimental): 1600 mg (two 800 mg in the form of tablets or powder to be diluted in water) TID with meals for 26 weeks
  Interventions: Drug: Sevelamer Carbonate
- calcium carbonate (Active Comparator): 1200 mg of calcium carbonate TID with meals for 26 weeks
  Interventions: Drug: calcium carbonate

INTERVENTIONS:
Drug: Sevelamer Carbonate — 1600 mg (two 800 mg in the form of tablets or powder to be diluted in water) TID with meals for 26 weeks
  Arms: Sevelamer Carbonate
Drug: calcium carbonate — 1200 mg of calcium carbonate TID with meals for 26 weeks
  Other Names: (Tums®)
  Arms: calcium carbonate

SUMMARY:
The purpose of this study is to see if taking a medication can lower the amount of oxidants from food that go into our body. Previous research shows that if the investigators lower the oxidants from food in people with diabetes, this simple change lowers different risks for heart disease and the worsening of kidney disease. The investigators focus on a specific type of oxidant, advanced glycation endproducts (AGEs). A previous, smaller study, conducted by our group showed that a drug, already approved by the FDA, will lower AGEs in the investigators compared Renvela® to Tums®. Both of these drugs have few side effects and have been used for a long time in patients with diabetes and kidney disease. While our previous study was interesting, it was just too small to be able to be sure that it will help all people with diabetes, or if the good effects the investigators found were simply due to chance. The investigators are doing this new study to confirm or deny the possibility that Renvela® can really help people with diabetes and kidney disease.

DETAILED DESCRIPTION:
Advanced glycation end products (AGEs) levels are elevated in diabetic patients and in patients with chronic kidney disease (CKD) and may contribute to the excessive cardiovascular disease in this population, by promoting oxidant stress and chronic vascular inflammation. It has recently been recognized that AGEs in the body originate not only endogenously, but also from the ingestion of preformed AGEs in the diet. We have shown that reduction of dietary AGE intake leads to significant reductions of circulating AGEs and insulin levels as well as levels of markers of oxidative stress and inflammation in both diabetic and CKD patients. Thus, the increased inflammation and oxidative stress (Infl/OS) in stable diabetes mellitus (DM) are largely due to advanced glycation end products (AGEs) from food, and restricting AGEs-intake reduces these risk factors in DM. High circulating AGEs and TNFR1/2 have been shown to be associated with progression in diabetic nephropathy. Ideally, a compound that binds food AGEs within the lumen of the intestine should have the same effect as dietary restriction of AGEs and could become an important therapeutic tool in the clinical care of these patients. We found that Sevelamer binds AGEs in vitro in a pH dependent manner. This led us to hypothesize that sevelamer carbonate, but not calcium carbonate, would sequester AGEs in the gut and reduce Infl/OS, including circulating AGEs and TNFα, in T2DM with Stage 2-4 CKD. This hypothesis was tested in a Pilot Study (GCO-08-0976) we designed as a proof-of-concept trial to determine if a larger and longer trial is indicated. We conducted a randomized, open-label, intention-to-treat, two-month crossover study to compare stable diabetic patients with stage 2-4 CKD treated with either Sevelamer carbonate or calcium carbonate for 2 months, a 1 week wash-out, and then the opposite drug for 2 months. There were no changes in medications and food intake. We found that urinary phosphate excretion was decreased by both Sevelamer carbonate and calcium carbonate. Serum AGEs, lipids, HbA1c, FGF23, and 8-isoprostanes were reduced by Sevelamer carbonate compared to calcium carbonate. In addition, PMNC levels of AGER1, SIRT1 and TNFα were also decreased by Sevelamer carbonate, compared to calcium carbonate. We concluded that Sevelamer carbonate reduces HbA1c, FGF23, lipids, and TNFα via reduced inflammation and OS in stage 2-4 diabetic CKD. These changes were not seen with calcium carbonate. Since we found that sevelamer carbonate bound AGE-BSA (but not BSA) at pH 7.0, but not at pH 1.0 in vitro, we proposed that the mechanism action is sequestration of dietary AGEs and GI elimination. Based on these data, we concluded that a larger and longer trial is indicated to confirm these results.

The current study proposes to confirm that Sevelamer Carbonate, an agent known to prevent the gastrointestinal absorption of phosphates, is also able to block the absorption of AGEs and improve certain aspects of diabetes and chronic renal disease in a larger group of patients who will be followed for a longer period of time.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Evidence of CKD Stages II, III or IV
* Stage II CKD; eGFR 60-89 ml/min
* Stage III CKD: eGFR 30-59 ml/min
* Stage IV CKD: eGFR 15-29 ml/min
* Proteinuria (>200 mg/day or 300 mg/gm creatinine on a spot urine) on urinalysis on two occasions within 18 months of recruitment
* Diagnosis of diabetes and receiving at least one medication for diabetes mellitus
* HbA1c>6.5%

Exclusion criteria:

* Age <18
* Patients receiving active treatment for hyperphosphatemia
* Biopsy proven renal disease other than diabetic nephropathy
* Hypophosphatemia
* Hypercalcemia
* Any history of significant gastrointestinal disorders
* Any history of significant gastrointestinal surgery such as ileostomy, colostomy and colectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
glucose metabolism | baseline
  HbA1C and serum AGE levels
glucose metabolism | at 3 months
  HbA1C and serum AGE levels
glucose metabolism | at 6 months
  HbA1C and serum AGE levels

SECONDARY OUTCOMES:
markers of inflammation and oxidative stress | baseline
markers of inflammation and oxidative stress | at 3 months
markers of inflammation and oxidative stress | at 6 months
serum lipid levels | baseline
serum lipid levels | at 3 months
serum lipid levels | at 6 months
serum phosphate level | at one week
  to check for hypophosphatemia
serum phosphate level | at two weeks
  to check for hypophosphatemia

CONTACTS AND LOCATIONS:
Overall Officials: Gary Striker, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Beth Israel Medical Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086
- [Derived] Vlassara H, Uribarri J, Cai W, Goodman S, Pyzik R, Post J, Grosjean F, Woodward M, Striker GE. Effects of sevelamer on HbA1c, inflammation, and advanced glycation end products in diabetic kidney disease. Clin J Am Soc Nephrol. 2012 Jun;7(6):934-42. doi: 10.2215/CJN.12891211. Epub 2012 Mar 29. PMID 22461535